CLINICAL TRIAL: NCT05717907
Title: Suction Catheter as a Guide for Nasotracheal Intubation Under General Anesthesia: Randomized Clinical Trial of Efficacy
Brief Title: Suction Catheter as a Guide for Nasotracheal Intubation Under General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Duangdee Rummasak, Assoc. Prof., Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023/DT039
Record Dates: First submitted 2023-01-16; First posted 2023-02-08 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Intubation Complication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): conventional nasotracheal intubation procedure
- Guided group (Experimental): use suction catheter guided endotracheal tube through the nasal passage
  Interventions: Device: suction catheter

INTERVENTIONS:
Device: suction catheter — a suction catheter will be first inserted through the ETT so that about 10 cm of the catheter was protruding from the distal end of the tube. The tip of the catheter is then inserted through the selected nostril until it passes to the pharynx. If resistance is felt to the passage of catheter, the other nostril will be tried. The nostril with less resistance to the catheter passage will be chosen for the completion of the procedure. The Endotracheal tube is then advance over the catheter through the nasal passage while holding the catheter proximal to the tube to prevent its advancement with the tube. After the tube tip reach to the pharynx, the suction catheter is withdrawn and tracheal intubation will be completed.
  Arms: Guided group

SUMMARY:
The goal of this clinical trial to study the efficacy of suction catheter guided technique and conventional technique during nasotracheal intubation.

The main question are

* How effective of the use of a suction catheter guided ETT in reducing bleeding during nasotracheal intubation?
* Does the use of a suction catheter guided ETT can improve its navigability through the nasal passage and reduce nasal passage time?

DETAILED DESCRIPTION:
Study design Clinical trial: Prospective randomized controlled trial with equal randomization (1:1), double-blinded (Participant and Primary outcome assessor), parallel design

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing elective oral and maxillofacial surgery in which nasotracheal intubation is preferred over orotracheal intubation to optimize surgical access.
* ASA physical status I-II
* Thai adult, aged 18-65 years old
* Normal Body Mass Index (BMI = 18.5-24.9)

Exclusion Criteria:

* Anticipated difficult airway (e.g., Mallampati classification 3-4, interincisal distance < 35 mm., thyromental length < 60 mm., limited neck mobility)
* Nasal infection or systemic infection
* Abnormal coagulation status or having bleeding disorder or taking anticoagulation/antiplatelet medication
* History of recurrent epistaxis since adulthood
* Allergic rhinitis that necessitates the use of glucocorticoids, antihistamine, antileukotriene or decongestant in the past 4 weeks
* History of nasal trauma or abnormality (e.g., trauma in mid-face region, nasal surgery, nasal polyps, chronic sinusitis, abnormal nasal vasculature, tumor in nasal region, radiotherapy in nasal region)
* Craniofacial deformity syndrome
* Using nasal oxygen or Continuous Positive Airway Pressure (CPAP)
* Previous nasotracheal intubation or nasogastric tube placement within 3 months
* Diagnosed as having a mental disorder

Drop-out criteria:

* Unable to complete intubation procedure
* Intubation failed on both nostrils
* When intubation was only possible with a tube smaller than 6.5 internal diameter (ID) in male and 6.0 ID in female
* Inadequate data collection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2024-06-09 (Actual); Study Completion 2024-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Duangdee Rummasak, M.D., Principal Investigator — Mahidol University
Locations (1):
- Faculty of Dentistry, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anwer HM.F., Ibrahim AA. Suction catheter guidance of the endotracheal tube to facilitate nasal intubation: a double blind, randomized clinical trial. MEJA.2018;25 (2):155-63.
- [Background] Prasanna D, Bhat S. Nasotracheal Intubation: An Overview. J Maxillofac Oral Surg. 2014 Dec;13(4):366-72. doi: 10.1007/s12663-013-0516-5. Epub 2013 May 1. PMID 26224998
- [Background] Jongcharoenkamon I, Juajarn T, Pisilp N. Does suction tube guiding reduce epistaxis from nasotracheal intubation? Mahasarakham Hospital Journal. 2020;17(3):210-7.
- [Background] Kim YC, Lee SH, Noh GJ, Cho SY, Yeom JH, Shin WJ, Lee DH, Ryu JS, Park YS, Cha KJ, Lee SC. Thermosoftening treatment of the nasotracheal tube before intubation can reduce epistaxis and nasal damage. Anesth Analg. 2000 Sep;91(3):698-701. doi: 10.1097/00000539-200009000-00038. PMID 10960403
- [Background] Piepho T, Thierbach A, Werner C. Nasotracheal intubation: look before you leap. Br J Anaesth. 2005 Jun;94(6):859-60. doi: 10.1093/bja/aei146. Epub 2005 Apr 15. PMID 15833776

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Guided Group
Started | 26 | 26
Completed | 26 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Guided Group | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (10) | 28.6 (10) | 29.8 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 11 | 10 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Mean (Standard Deviation); unit: kilograms] | 59.5 (10.3) | 60 (10.8) | 59.8 (10.5)
Height [Mean (Standard Deviation); unit: centimetres] | 165.3 (8.7) | 167.3 (10.1) | 166.3 (9.4)
ASA physical status [Count of Participants; unit: Participants] — ASA I; normal healthy ASA II; mild systemic disease controllable
  Participants
    I | 21 | 22 | 43
    II | 5 | 4 | 9
Type of Diagnosis [Count of Participants; unit: Participants]
  Dentofacial deformities | 19 | 21 | 40
  Pathology | 3 | 2 | 5
  Miscellaneous | 4 | 3 | 7
Type of operation [Count of Participants; unit: Participants]
  Orthognathic and/or adjunctive surgery | 19 | 21 | 40
  Excision and/or reconstruction | 4 | 2 | 6
  Minor dentoalveolar surgery | 3 | 3 | 6
History of smoking [Count of Participants; unit: Participants]
  Never | 22 | 23 | 45
  Cessation | 3 | 2 | 5
  Current | 1 | 1 | 2
History of alcohol consumption [Count of Participants; unit: Participants]
  Never | 18 | 14 | 32
  Occasional (<1 time/week) | 7 | 11 | 18
  Regular (more than 1 time/week) | 1 | 1 | 2
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 14 (1.3) | 13.8 (1.4) | 13.9 (1.3)
Platelet count [Mean (Standard Deviation); unit: platelets/microlitre] — *1000/microliter
  platelets/microlitre | 291000 (60000.9) | 271200 (64500) | 281100 (62900)
Mean arterial pressure (MAP) [Mean (Standard Deviation); unit: mmHg] | 89 (9) | 88 (11) | 88 (10)
Nostril selected by patient [Count of Participants; unit: Participants]
  Right | 12 | 12 | 24
  Left | 9 | 8 | 17
  Undecided | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Extent of Bleeding
Description: The video from video laryngoscope will be recorded at the moment during and immediately after successful intubation, which will be later reviewed by primary outcome assessor that not involved in the procedure. Accounting for only bleeding observed at posterior pharyngeal area, which originate from trauma from attempt to pass ETT through the nasal passage into the pharynx. Assessment of bleeding will be scored at the most severe bleeding state observed from inserting to the removal of video laryngoscope after successful intubation. The extent of bleeding will be graded as:
  "Grade 0" = no bleeding "Grade 1" = blood-stained tube and/or cuff "Grade 2" = blood-stained posterior pharyngeal wall (traces or streak of blood) "Grade 3" = blood pooling at posterior pharyngeal wall
Time Frame: measured from video recorded at insert to withdraw videolaryngoscope
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Guided Group
Number analyzed (Participants) | 26 | 26
Participants
  Grade 0 | 12 | 13
  Grade 1 | 3 | 3
  Grade 2 | 4 | 3
  Grade 3 | 7 | 7
Statistical Analysis 1: Comparison: Control Group vs Guided Group; Test type: Superiority; p = 1.000, Chi-squared

2. Primary Outcome: Incidence of Bleeding
Description: rate of incidence of bleeding
  * No Bleeding (Grade 0)
  * Bleeding (Grade 1, 2, 3)
Time Frame: measured immediately after successful intubation
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Guided Group
Number analyzed (Participants) | 26 | 26
Participants
  No bleeding | 12 | 13
  Bleeding | 14 | 13

3. Secondary Outcome: Ease of Navigation
Description: Ease of navigation during advancement of tube though the nasal passage, will be recorded as "Smooth" = ETT meet no resistance, no need to adjust the tube "Slight resistance" = ETT meet the resistance and has to be manipulated more than once "Impinged" = ETT cannot pass through and need to move to another nostril
Time Frame: measured immediately after successful intubation
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Guided Group
Number analyzed (Participants) | 26 | 26
Participants
  Smooth | 20 | 22
  Slight resistance | 2 | 3
  Impinged | 4 | 1

4. Other Pre Specified Outcome: Number of Attempts
Description: The outcome will be recorded as "1,2,3,...." Number of insertion attempt to pass the nasal passage in each participants.
Time Frame: measured immediately after successful intubation
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Guided Group
Number analyzed (Participants) | 26 | 26
Participants
  1 | 22 | 25
  2 | 2 | 0
  3 | 1 | 1
  6 | 1 | 0

5. Other Pre Specified Outcome: Nasal Passage Time
Description: * Control group: starting when the tip of the ETT just enter the anterior nares until the tip of the ETT just pass the posterior nares and entered the pharynx
  * Guided group: starting when the tip of the guiding suction catheter just entered the anterior nares until the tip of the ETT passed the posterior nares, then entered the pharynx and the guiding catheter was completely removed from the ETT.
  The outcome will be recorded in "unit of seconds"
Time Frame: measured immediately after successful intubation
Measure: Median (Full Range); unit: seconds
Arm/Group | Control Group | Guided Group
Number analyzed (Participants) | 26 | 26
seconds | 5.4 [3.1 to 67.5] | 10.3 [6.0 to 42.2]

ADVERSE EVENTS:
Time Frame: 1 hr after extubation
Description: * inability to complete intubation process
  * Major bleeding events
  * False tract/ mucosal laceration
  * Turbinectomy
Arm/Group | Control Group | Guided Group
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-11): https://cdn.clinicaltrials.gov/large-docs/07/NCT05717907/Prot_SAP_000.pdf